CLINICAL TRIAL: NCT02675894
Title: Switching Bipolar Radiofrequency Ablation Using Cooled-Wet Electrode for Treatment of Hepatocellular Carcinoma: A Preliminary Study
Brief Title: Radiofrequency Ablation Using Cooled-Wet Electrode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: RF medical (Unknown); Medical Research Collaborating Center (Unknown)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNUH-2013-2283
Record Dates: First submitted 2016-02-01; First posted 2016-02-05 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: HCC; Metastasis
Keywords: RFA
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA with cooled-wet electrode (Active Comparator): RFA is performed using three cool-wet electrodes in switching bipolar mode under the fused US guidance.
  Interventions: Device: cooled-wet electrode
- RFA with separable clustered electrode (Active Comparator): RFA using separable clustered electrode in switching monopolar mode under the fused US guidance
  Interventions: Device: separable clustered electrode

INTERVENTIONS:
Device: cooled-wet electrode — RFA is performed using three cooled-wet electrodes in switching bipolar mode. The electrode is anticipated to reduce tissue resistance by releasing small amount of saline during the procedure, which may lead larger ablative volume by delivering more RF energy.
  Arms: RFA with cooled-wet electrode
Device: separable clustered electrode — RFA is performed using separable clustered electrode in switching monopolar mode.
  Other Names: Octopus(R)
  Arms: RFA with separable clustered electrode

SUMMARY:
To determine safety, ablative zone, technical success rate and early safety data of recently introduced cool-wet electrode in eligible patients who are indicative for radiofrequency ablation (RFA) for liver tumors.

DETAILED DESCRIPTION:
To determine safety, ablative zone, technical success rate and early safety data (12 months local tumor progression rate) of recently introduced cooled-wet electrode in eligible patients who are indicative for radiofrequency ablation (RFA) for liver tumors in comparison with currently used separable clustered electrode in our institution. Owing to tissue cooling effect of internally cooled-wet electrode can be used in switching bipolar mode. Patients would be randomized into two groups (cool-wet electrode group and separable clustered electrode in switching monopolar mode). The results from this preliminary study would be used for main study to compare the efficacy and safety data between two electrodes in the future.

ELIGIBILITY:
Inclusion Criteria: all conditions have to be fulfilled.

* Diagnosed with HCC (1~5cm) according to AASLD guideline or LI-RADS on MDCT or liver MRI within 60 days before RFA
* liver metastasis histologically confirmed or characteristic findings on cross-sectional imaging
* signed informed consent
* treatment naive index tumor (no history of local treatment for an index tumor)

Exclusion Criteria:

* more than three tumors in a patients
* tumor size larger than 5cm
* tumor attaches to central portal vein or hepatic vein
* Child-Pugh classification C
* uncorrected coagulopathy
* presence of extrahepatic metastases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
LTP | 24 months
  cumulating local tumor progression rate over 2- year after RFA

SECONDARY OUTCOMES:
Technical success rate | 1 months
  technical success rate on 1 month follow-up which indicates no residual tumor on cross-sectional imaging (CT, MRI)
IDR rate | 24 months
  cumulating intrahepatic distant recurrence (IDR) rate over 2- year after RFA
EM rate | 24 months
  cumulating extrahepatic metastasis (EM) rate over 2- year after RFA
Maximal diameter of ablative zone | 7 day
  Maximal diameter of ablative zone on post-RFA CT or MRI in a mm.
ablation time | 1 day
  RFA procedure time in each patient.
Complication | 12 months
  all complication rate and grades (according to Clavien system from I to III) related with RFA procedure
Volume of ablative zone | 7 days
  Volume of ablative zone on post-RFA CT or MRI in a mm3.

OTHER OUTCOMES:
US/CT or MR fusion success rate | 1 day
  RFA is performed under real time US guidance and US is fused with pre-RFA CT or MRI before ablation of the index tumor. US/CT or US/MR fusion quality is assessed by an operator.
Immediate assess of technique success rate | 2 days
  After performing RFA, patients were transferred CT unit to confirm immediate technique success. It is performed in both a) visual inspection using pre-and post-RFA images side-by-side comparison and b) software assisted inspection which register pre-and post-RFA scans. The results would be used to perform additional treatment (2nd look RFA).

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No